CLINICAL TRIAL: NCT00223132
Title: Suture Granuloma in Body Contouring Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: SYN04002
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Skin Laxity of Abdomen, Thighs, Chest, Back, and Neck
Keywords: bariatric surgery; body contouring; skin laxity; plastic surgery; suture granuloma; absorbable sutures
MeSH Terms: conditions — Cutis Laxa

INTERVENTIONS:
Device: Absorbable sutures

SUMMARY:
The purpose of this study is to evaluate the effect of different suture material on the incidence of suture granuloma.

DETAILED DESCRIPTION:
Bariatric surgery has evolved as an effective treatment for morbid obesity, inducing rapid and predictable weight loss within a period of 12 to 18 months following surgery. Consequently, body contouring after weight loss is emerging as the fastest growing field of plastic surgery. Patients seek consultation with a plastic surgeon to correct skin laxity of the abdomen, thighs, chest, back, and neck.

A major problem in body contourinig is the extrusion of absorbable suture material used for dermal closure. Long incisions and high tension inherent to body contouring surgery mandate a secure dermal closure. While absorbable sutures are preferred, they can result in suture granuloma and extrusion.

ELIGIBILITY:
Inclusion Criteria:

Men and women 18 years and older

Exclusion Criteria:

Subjects with active infectious collagen disease,significant anatomic asymmetry that creates markedly different wound tension and/or geometry between left and right side Subjects who cancel their surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Doran, Study Director — Medtronic - MITG
Locations (1):
- University Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States